CLINICAL TRIAL: NCT01101022
Title: A Phase 4, Randomized, Double-Blind, Multicenter, Placebo-controlled, Parallel Group Study Evaluating the Safety and Efficacy of SPD489 on Executive Function (Self-Regulation) Behaviors in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD) Reporting Clinically Significant Impairment of Real-World Executive Function Behavior.
Brief Title: Safety and Efficacy of SPD489 on Executive Function Behaviors in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-403
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Results first posted 2012-02-13 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: ADHD Specifically With Executive Function Impairment
MeSH Terms: interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPD489 (Active Comparator)
  Interventions: Drug: SPD489
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SPD489 — 1 capsule per day (30, 50 or 70 mg), daily throughout the double-blind treatment period (10 weeks)
  Other Names: Vyvanse
  Arms: SPD489
Other: Placebo — 1 capsule per day, daily throughout the double-blind treatment period (10 weeks)
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of SPD489 compared to placebo on executive function (self-regulation) behaviors in adults with ADHD who report clinically significant impairment of executive function behavior in their everyday environment, as measured by the self-report Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A) Global Executive Composite (GEC) T-score.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18-55 years of age, inclusive at the time of consent.
2. Subject has an established close relationship of at least 6-months duration before screening (Visit -1) with an informant who will be able to observe and be willing to report on the subject's behavior and symptoms in multiple social settings during the course of the study. Informant is defined as a person who has a domicile relationship with the subject. When applicable, the informant should be the subject's spouse/significant other. Additionally, the informant cannot participate as a subject in the study and can only serve as the informant for a single subject.
3. Subject has a lifestyle that in the opinion of the Investigator will enable the subject to complete all study testing and requirements defined in the protocol.
4. Female subjects must have a negative serum beta human chorionic gonadotropin (HCG) pregnancy test at screening (Visit -1) and a negative urine pregnancy test at baseline (Visit 0) and agree to comply with any applicable contraceptive requirements of the protocol.
5. Subject meets the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM-IV-TR) criteria for a primary diagnosis of ADHD (diagnostic code 314.00 and 314.01) established by a comprehensive psychiatric evaluation that reviews DSM-IV-TR criteria with at least 6 of the 9 subtype criteria met. The Adult ADHD Clinical Diagnostic Scale version 1.2 (ACDS v1.2) will be utilized as the diagnostic tool.
6. Subject has a total score of ≥65 on BRIEF-A GEC T-score by self-report at baseline (Visit 0).
7. Subject has a total score of ≥28 using the Adult ADHD-RS with prompts at baseline (Visit 0).
8. Subject must have a minimum level of intellectual functioning as determined by the Investigator at screening (Visit -1).
9. Subject is able to swallow a capsule.
10. Subject is willing and able to comply with all the testing and requirements defined in this protocol.
11. Subject and informant must be able to provide written, personally signed and dated informed consent to participate in the study in accordance with the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guidelines and applicable regulations before completing any study related procedures.

Exclusion Criteria

1. Subject has a current comorbid psychiatric disorder that is either controlled with medications prohibited in this study or is uncontrolled and associated with significant symptoms. Prohibited disorders include those associated with diagnoses including but not limited to any severe comorbid Axis II disorder or severe Axis I disorder (such as Post Traumatic Stress Disorder [PTSD], psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder). Other symptomatic manifestations (such as agitated states) that contraindicate treatment with SPD489 or confound efficacy or safety assessments in the opinion of the examining physician are also prohibited. Comorbid psychiatric diagnoses will be established by the psychiatric evaluation that includes the Structured Clinical Interview for DSM-IV-TR disorders (SCID-I).
2. Subjects who are currently considered a suicide risk, any subject who has previously made a suicide attempt or those who are currently demonstrating active suicidal ideation.
3. The subject has a body mass index (BMI) of <18.5 or ≥40.
4. Subject has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might confound the results of safety assessments administered in the study or that might increase risk to the subject. Similarly, the subject will be excluded if he or she has any additional condition(s) that in the Investigator's opinion would prohibit the subject from completing the study or would not be in the best interest of the subject. This would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol. Mild, stable asthma is not exclusionary.
5. Subject has a history of seizures (other than infantile febrile seizures), any tic disorder, a current diagnosis and/or a known family history of Tourette's Disorder.
6. Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, transient ischemic attack or stroke or other serious cardiac problems that may place them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
7. Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
8. Subject has any clinically significant ECG or clinically significant laboratory abnormality at screening (Visit -1).
9. Subject has current abnormal thyroid function, defined as abnormal screening thyroid stimulating hormone (TSH) and thyroxine (T4). Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
10. Subject has a history of moderate to severe hypertension or has a resting sitting systolic blood pressure >139mmHg or diastolic blood pressure >89mmHg. Subjects with well-controlled mild or moderate hypertension on a single antihypertensive agent are allowed. Combination antihypertensive medications are not allowed.
11. Subject is taking any medication that is excluded.
12. Subject has a documented allergy, hypersensitivity, or intolerance to amphetamines.
13. Subject has a documented allergy, hypersensitivity, or intolerance to any excipients in the investigational medicinal product.
14. Subject has failed to respond to one or more adequate courses (dose and duration) of amphetamine therapy.
15. Subject has a recent history (within the past 6 months) of suspected substance abuse or dependence disorder (excluding nicotine) in accordance with DSM-IV-TR criteria.
16. Subject has a positive urine drug result at screening (Visit -1) (with the exception of subject's current stimulant therapy, if any).
17. Subject has taken an investigational drug or taken part in a clinical trial, including an SPD489 clinical trial, within 30 days prior to screening (Visit -1).
18. Subject has glaucoma.
19. Subject is taking other medications that have central nervous system (CNS) effects or affect performance, such as sedating antihistamines and decongestant sympathomimetics, or are monoamine oxidase inhibitors (during or within 7 days of investigational medicinal product administration). Stable use of bronchodilator inhalers is not exclusionary.
20. Subject is female and pregnant or lactating.
21. Subjects who have previously been randomized into this study and subsequently withdrawn.
22. Subject is well controlled on their current ADHD medication with acceptable tolerability.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2010-05-19 (Actual); Primary Completion 2010-11-29 (Actual); Study Completion 2010-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (39):
- United States (39):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Peninsula Research Assoc, Inc, Rolling Hills Estates, California
  - PCSD Feighner Research, San Diego, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Dr. George Joseph, MD and Associates PA, Jacksonville Beach, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - CNS Healthcare, Orlando, Florida
  - Janus Center For Psychiatric Research, West Palm Beach, Florida
  - Atlanta Center For Medical Research, Atlanta, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - AMR-BABER Research Inc., Naperville, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - Vince and Associates Clinical Research, Inc., Overland Park, Kansas
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Mark Hertzman MD, PC, Rockville, Maryland
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - The Behavioral Medicine Clinic of NW Michigan, PC, Traverse City, Michigan
  - Midwest Research Group, Saint Charles, Missouri
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Bioscience Research, LLC, Mount Kisco, New York
  - Mental Health and Addictive Disorders Research Program, New York, New York
  - Triangle Neuropsychiatry, Durham, North Carolina
  - Richard H. Weisler, MD, Pa & Associates, Raleigh, North Carolina
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Occi, Inc (Oregon Center For Clinical Investigations, Inc.), Salem, Oregon
  - FutureSearch Trials, LP, Austin, Texas
  - Bayou City Research, Ltd., Houston, Texas
  - Red Oak Psychiatry Associates P.A., Houston, Texas
  - John M. Turnbow, MD, PA, Lubbock, Texas
  - Vermont Clinical Study Center, Burlington, Vermont
  - Neuropsychiatric Associates, Woodstock, Vermont
  - Neuroscience, Inc, Herndon, Virginia
  - Eastside Therapeutic Resource, Kirkland, Washington
  - Summit Research Network, LLC, Seattle, Washington
  - Rockwood Clinic, Spokane, Washington
  - Dean Foundation for Health, Research and Education, Middleton, Wisconsin

REFERENCES:
- [Result] Adler LA, Dirks B, Deas PF, Raychaudhuri A, Dauphin MR, Lasser RA, Weisler RH. Lisdexamfetamine dimesylate in adults with attention-deficit/ hyperactivity disorder who report clinically significant impairment in executive function: results from a randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2013 Jul;74(7):694-702. doi: 10.4088/JCP.12m08144. PMID 23945447
- [Derived] Brown TE, Chen J, Robertson B. Relationships Between Executive Function Improvement and ADHD Symptom Improvement With Lisdexamfetamine Dimesylate in Adults With ADHD and Executive Function Deficits: A Post Hoc Analysis. Prim Care Companion CNS Disord. 2020 May 28;22(3):19m02559. doi: 10.4088/PCC.19m02559. PMID 32470230
- [Derived] Adler LA, Dirks B, Deas P, Raychaudhuri A, Dauphin M, Saylor K, Weisler R. Self-Reported quality of life in adults with attention-deficit/hyperactivity disorder and executive function impairment treated with lisdexamfetamine dimesylate: a randomized, double-blind, multicenter, placebo-controlled, parallel-group study. BMC Psychiatry. 2013 Oct 9;13:253. doi: 10.1186/1471-244X-13-253. PMID 24106804

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 161 subjects were enrolled and randomized, but 2 never received any investigational product, and therefore were not included in subject disposition going forward (n = 159).
Groups:
- SPD489: Dosed orally once a day at approximately 7:00 AM at either 30, 50 or 70 mg for 10 weeks (a 4-week dose optimization period followed by a 6-week dose maintenance period at an optimal dose).
- Placebo: Dosed orally once a day at approximately 7:00 AM for 10 weeks.
Period: Overall Study
Arm/Group | SPD489 | Placebo
Started | 79 | 80
Completed | 62 | 53
Not Completed | 17 | 27
Not completed — Adverse Event | 6 | 2
Not completed — Protocol Violation | 4 | 3
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Lost to Follow-up | 1 | 4
Not completed — Lack of Efficacy | 0 | 7
Not completed — Sponsor decision | 1 | 1
Not completed — Non-compliance | 1 | 0
Not completed — Work schedule | 1 | 1
Not completed — Vacation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD489 | Placebo | Total
Number analyzed (Participants) | 79 | 80 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (10.58) | 34.9 (11.02) | 34.6 (10.77)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  18 to 55 years | 79 | 80 | 159
  >55 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 76
  Male | 40 | 43 | 83
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 79 | 80 | 159

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Subject-reported Behavior Rating Inventory of Executive Function - Adult Version Global Executive Composite T-score (BRIEF-A GEC T) at up to 10 Weeks
Description: BRIEF-A Global Executive Composite assesses behavioral aspects of executive function. Items are rated 1 (never), 2 (sometimes), and 3 (often). There is no range for a total score. Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline and up to 10 weeks
Population: Full Analysis Set (FAS) defined as all subjects who took 1 dose of investigational product in the double-blind evaluation phase and had 1 primary efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 79 | 75
T-scores | -22.3 (1.67) | -11.1 (1.72)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -11.2, 95% CI 2-sided [-15.9 to -6.4]

2. Secondary Outcome: Change From Baseline in Adult ADHD Impact Module (AIM-A) Multi-Item Scales Total Score at up to 10 Weeks
Description: The AIM-A was developed to assess impact of core ADHD symptoms on daily functioning and quality of life. For multi-item scales, subjects respond to items using a Likert scale with responses ranging from 1 (strongly agree) to 5 (strongly disagree). Scores were computed by deriving the mean of the item sets and transforming the scale score on a continuum from 0 to 100 using a standard formula. Higher scores indicate a better quality of life.
Time Frame: Baseline and up to 10 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 79 | 75
Scores on a scale
  Performance and Daily Functioning | 38.8 (2.84) | 17.2 (2.91)
  Impact of symptoms: Daily Interference | 30.6 (2.52) | 15.7 (2.58)
  Impact of symptoms: Bother/Concern | 29.3 (2.53) | 15.8 (2.60)
  Relationships/Communication | 21.2 (2.49) | 13.4 (2.56)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Performance and Daily Functioning; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 21.6, 95% CI 2-sided [13.5 to 29.7]
Statistical Analysis 2: Comparison: SPD489 vs Placebo; Daily Interference; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 14.9, 95% CI 2-sided [7.8 to 22.0]
Statistical Analysis 3: Comparison: SPD489 vs Placebo; Bother/Concern; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Final Values) = 13.5, 95% CI 2-sided [6.3 to 20.7]
Statistical Analysis 4: Comparison: SPD489 vs Placebo; Relationships/Communication; Test type: Superiority or Other; p = 0.0302, ANCOVA; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [0.8 to 14.9]

3. Secondary Outcome: Change From Baseline in Informant-reported BRIEF-A T-scores at up to 10 Weeks
Description: BRIEF-A is a validated 75-item questionnaire composed of three indexes (Global Executive Composite, Behavioral Recognition Index, and Metacognition Index). Items are rated 1 (never), 2 (sometimes), and 3 (often). Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline and up to10 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 71 | 71
T-scores
  Global Executive Composite | -10.2 (1.06) | -5.3 (1.06)
  Behavioral Regulation Index | -8.6 (1.04) | -5.5 (1.04)
  Metacognition Index | -10.3 (1.07) | -4.6 (1.07)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Global Executive Composite; Test type: Superiority or Other; p = 0.0016, ANCOVA; Mean Difference (Final Values) = -4.9, 95% CI 2-sided [-7.8 to -1.9]
Statistical Analysis 2: Comparison: SPD489 vs Placebo; Behavioral Regulation Index; Test type: Superiority or Other; p = 0.0355, ANCOVA; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-6.0 to -0.2]
Statistical Analysis 3: Comparison: SPD489 vs Placebo; Metacognition Index; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-8.7 to -2.7]

4. Secondary Outcome: Change From Baseline in Subject-reported BRIEF-A T-scores at up to 10 Weeks
Description: BRIEF-A is a validated 75-item questionnaire composed of three indexes (Global Executive Composite, Behavioral Recognition Index, and Metacognition Index). Global Executive Composite was reported as the Primary Outcome. Items are rated 1 (never), 2 (sometimes), and 3 (often). There is no range for a total score. Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline and up to 10 weeks
Population: FAS
Measure: Mean (Standard Error); unit: T-scores
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 79 | 75
T-scores
  Behavioral Regulation Index | -17.5 (1.54) | -9.2 (1.58)
  Metacognition Index | -22.8 (1.63) | -11.2 (1.67)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Behavioral Regulation Index; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -8.4, 95% CI 2-sided [-12.7 to -4.0]
Statistical Analysis 2: Comparison: SPD489 vs Placebo; Metacognition Index; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -11.6, 95% CI 2-sided [-16.3 to -7.0]

5. Secondary Outcome: Change From Baseline in Subject-reported BRIEF-A Clinical Subscales T-scores at up to 10 Weeks
Description: BRIEF-A clinical subscales items are rated 1 (never), 2 (sometimes), and 3 (often). There is no range for a total score. Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline and up to 10 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 79 | 75
T-scores
  Inhibit | -17.8 (1.50) | -9.5 (1.54)
  Shift | -14.5 (1.46) | -7.8 (1.50)
  Emotional control | -10.9 (1.28) | -5.7 (1.31)
  Self-monitor | -16.6 (1.44) | -8.4 (1.48)
  Initiate | -17.9 (1.38) | -8.6 (1.41)
  Working memory | -23.2 (1.67) | -11.9 (1.71)
  Plan/Organize | -20.8 (1.58) | -9.9 (1.62)
  Task monitor | -20.1 (1.64) | -10.8 (1.68)
  Organization of materials | -16.5 (1.26) | -7.6 (1.30)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Inhibit; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -8.3, 95% CI 2-sided [-12.6 to -4.1]
Statistical Analysis 2: Comparison: SPD489 vs Placebo; Shift; Test type: Superiority or Other; p = 0.0018, ANCOVA; Mean Difference (Final Values) = -6.7, 95% CI 2-sided [-10.8 to -2.5]
Statistical Analysis 3: Comparison: SPD489 vs Placebo; Emotional control; Test type: Superiority or Other; p = 0.0056, ANCOVA; Mean Difference (Final Values) = -5.2, 95% CI 2-sided [-8.8 to -1.5]
Statistical Analysis 4: Comparison: SPD489 vs Placebo; Sef-monitor; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -8.2, 95% CI 2-sided [-12.3 to -4.1]
Statistical Analysis 5: Comparison: SPD489 vs Placebo; Initiate; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -9.3, 95% CI 2-sided [-13.2 to -5.4]
Statistical Analysis 6: Comparison: SPD489 vs Placebo; Working memory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -11.3, 95% CI 2-sided [-16.0 to -6.6]
Statistical Analysis 7: Comparison: SPD489 vs Placebo; Plan/Organize; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -10.9, 95% CI 2-sided [-15.4 to -6.4]
Statistical Analysis 8: Comparison: SPD489 vs Placebo; Task monitor; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -9.3, 95% CI 2-sided [-14.0 to -4.7]
Statistical Analysis 9: Comparison: SPD489 vs Placebo; Organization of materials; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -8.9, 95% CI 2-sided [-12.5 to -5.3]

6. Secondary Outcome: Change From Baseline in Informant-reported BRIEF-A Clinical Subscales T-scores at up to 10 Weeks
Description: as for outcome 5
Time Frame: Baseline and up to 10 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 71 | 71
T-scores
  Inhibit | -10.2 (1.08) | -5.8 (1.08)
  Shift | -9.1 (1.17) | -4.3 (1.17)
  Emotional control | -5.9 (0.99) | -4.6 (0.99)
  Self-monitor | -6.8 (1.04) | -4.6 (1.04)
  Initiate | -8.6 (1.00) | -3.2 (1.00)
  Working memory | -12.0 (1.22) | -5.7 (1.22)
  Plan/Organize | -9.9 (1.07) | -5.0 (1.07)
  Task monitor | -9.7 (1.21) | -3.4 (1.21)
  Organization of materials | -6.2 (0.97) | -3.0 (0.97)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Inhibit; Test type: Superiority or Other; p = 0.0048, ANCOVA; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-7.4 to -1.4]
Statistical Analysis 2: Comparison: SPD489 vs Placebo; Shift; Test type: Superiority or Other; p = 0.0045, ANCOVA; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-8.0 to -1.5]
Statistical Analysis 3: Comparison: SPD489 vs Placebo; Emotional control; Test type: Superiority or Other; p = 0.3605, ANCOVA; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-4.0 to 1.5]
Statistical Analysis 4: Comparison: SPD489 vs Placebo; Self-monitor; Test type: Superiority or Other; p = 0.1468, ANCOVA; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-5.1 to 0.8]
Statistical Analysis 5: Comparison: SPD489 vs Placebo; Initiate; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -5.5, 95% CI 2-sided [-8.3 to -2.7]
Statistical Analysis 6: Comparison: SPD489 vs Placebo; Working memory; Test type: Superiority or Other; p = 0.0004, ANCOVA; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-9.8 to -2.9]
Statistical Analysis 7: Comparison: SPD489 vs Placebo; Plan/Organize; Test type: Superiority or Other; p = 0.0015, ANCOVA; Mean Difference (Final Values) = -4.9, 95% CI 2-sided [-7.9 to -1.9]
Statistical Analysis 8: Comparison: SPD489 vs Placebo; Task monitor; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-9.7 to -2.9]
Statistical Analysis 9: Comparison: SPD489 vs Placebo; Organization of materials; Test type: Superiority or Other; p = 0.0234, ANCOVA; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-5.9 to -0.4]

7. Secondary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) With Adult Prompts Total Score at up to 10 Weeks
Description: The ADHD-RS consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54. Lower scores indicate reduction in symptoms.
Time Frame: Baseline and up to 10 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 79 | 75
Scores on a scale | -21.4 (1.35) | -10.3 (1.38)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -11.1, 95% CI 2-sided [-14.9 to -7.3]

8. Secondary Outcome: Percent of Participants With Clinical Global Impression - Severity of Illness (CGI-S) at Baseline
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill)
Time Frame: Baseline
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 79 | 75
Percent of participants
  Normal, not at all ill | 0 | 0
  Borderline mentally ill | 0 | 0
  Mildly ill | 0 | 0
  Moderately ill | 48.1 | 42.7
  Markedly ill | 38.0 | 49.3
  Severely ill | 13.9 | 8.0
  Among the most extremely ill | 0 | 0

9. Secondary Outcome: Percent of Participants With Clinical Global Impression - Severity of Illness (CGI-S) at up to 10 Weeks
Description: as for outcome 8
Time Frame: Up to 10 weeks post-dose
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 79 | 75
Percent of participants
  Normal, not at all ill | 13.9 | 6.7
  Borderline mentally ill | 38.0 | 16.0
  Mildly ill | 21.5 | 10.7
  Moderately ill | 15.2 | 37.3
  Markedly ill | 8.9 | 25.3
  Severely ill | 2.5 | 4.0
  Among the most extremely ill | 0 | 0

10. Secondary Outcome: Percent of Participants With Improvement on Clinical Global Impression - Global Improvement (CGI-I) at up to 10 Weeks
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: Up to 10 weeks post-dose
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 79 | 75
Percent of participants | 78.5 | 34.7
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared

11. Secondary Outcome: Change From Baseline in AIM-A Multi-Item Scales of Living With ADHD and General Well-being Score at up to 10 Weeks
Description: as for outcome 2
Time Frame: Baseline and up to 10 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 79 | 75
Scores on a scale
  Living with ADHD | 14.0 (1.30) | 4.9 (1.33)
  General Well-being | 19.7 (1.69) | 9.0 (1.73)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Living with ADHD; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 9.1, 95% CI 2-sided [5.4 to 12.7]
Statistical Analysis 2: Comparison: SPD489 vs Placebo; General Well-being; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 10.8, 95% CI 2-sided [6.0 to 15.5]

12. Secondary Outcome: Change From Baseline in AIM-A Quality of Life Questions 1 and 4 Scores at up to 10 Weeks
Description: Question 1: 'On a scale of 1 to 10, how would you rate the overall quality of life right now?' It is rated on a scale of 1 (worst) to 10 (best). Higher scores representing a more positive rating. Question 4: 'How much do you agree with this statement: Over the past few weeks, I've had more good days than bad days?' This is rated on a scale of 1 (strongly agree) to 5 (strongly disagree). Lower scores represent better quality of life.
Time Frame: Baseline and up to 10 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 79 | 75
Scores on a scale
  Question 1 | 1.6 (0.16) | 1.0 (0.16)
  Question 4 | -1.0 (0.11) | -0.4 (0.11)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Question 1; Test type: Superiority or Other; p = 0.0184, ANCOVA; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [0.1 to 1.0]
Statistical Analysis 2: Comparison: SPD489 vs Placebo; Question 4; Test type: Superiority or Other; p = 0.0004, ANCOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.9 to -0.3]

13. Secondary Outcome: Change From Baseline in Conner's Adult ADHD Rating Scale-Observer: Short Version (CAARS-O:S) ADHD Index T-score at up to 10 Weeks
Description: The CAARS-O:S is an assessment tool with prompts provided to an observer who describes ADHD-related symptoms in an adult subject. The 26-item scale is scored on a 4-point scale from 0 (not at all) to 3 (very much, very frequently). There is no range for a total score. Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline and up to 10 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 71 | 71
T-scores | -11.3 (1.24) | -5.8 (1.24)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Test type: Superiority or Other; p = 0.0019, ANCOVA; Mean Difference (Final Values) = -5.5, 95% CI 2-sided [-9.0 to -2.1]

14. Secondary Outcome: Change From Baseline in CAARS-O:S Factor-derived Subscale T-scores at up to 10 Weeks
Description: as for outcome 13
Time Frame: Baseline and up to 10 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 71 | 71
T-scores
  Inattention/Memory Problems | -10.0 (1.12) | -4.9 (1.12)
  Hyperactivity/Restlessness | -9.1 (1.20) | -5.0 (1.20)
  Impulsivity/Emotional Liability | -8.0 (1.01) | -4.0 (1.01)
  Problems with Self-concept | -7.7 (1.10) | -3.3 (1.10)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Inattention/Memory Problems; Test type: Superiority or Other; p = 0.0017, ANCOVA; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-8.2 to -1.9]
Statistical Analysis 2: Comparison: SPD489 vs Placebo; Hyperactivity/Restlessness; Test type: Superiority or Other; p = 0.0174, ANCOVA; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-7.5 to -0.7]
Statistical Analysis 3: Comparison: SPD489 vs Placebo; Impulsivity/Emotional Liability; Test type: Superiority or Other; p = 0.0063, ANCOVA; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-6.8 to -1.1]
Statistical Analysis 4: Comparison: SPD489 vs Placebo; Problems with Self-concept; Test type: Superiority or Other; p = 0.0059, ANCOVA; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-7.5 to -1.3]

15. Secondary Outcome: Change From Baseline in Adult ADHD Quality of Life (AAQoL) Scale Total Score at up to 10 Weeks
Description: AAQoL is a validated 29-item scale consisting of 4 subscales. The AAQoL yields a total score and 4 subscale scores. Subjects rate each item on a 5-point Likert scale ranging from 1 (not at all/never) to 5 (extremely/very often). These scores are then transformed to a 0-100 point scale with higher scores indicating better quality of life.
Time Frame: Baseline and up to 10 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 28 | 26
Scores on a scale
  Life Productivity | 38.0 (4.34) | 17.0 (4.51)
  Psychological Health | 19.3 (3.61) | 7.2 (3.74)
  Life Outlook | 18.5 (2.85) | 6.0 (2.96)
  Relationships | 17.1 (3.69) | 9.8 (3.83)
  Total Score | 25.9 (3.04) | 11.1 (3.16)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Life Productivity; Test type: Superiority or Other; p = 0.0016, ANCOVA; Mean Difference (Final Values) = 21.0, 95% CI 2-sided [8.4 to 33.6]
Statistical Analysis 2: Comparison: SPD489 vs Placebo; Psychological Health; Test type: Superiority or Other; p = 0.0242, ANCOVA; Mean Difference (Final Values) = 12.1, 95% CI 2-sided [1.6 to 22.5]
Statistical Analysis 3: Comparison: SPD489 vs Placebo; Life Outlook; Test type: Superiority or Other; p = 0.0038, ANCOVA; Mean Difference (Final Values) = 12.5, 95% CI 2-sided [4.2 to 20.8]
Statistical Analysis 4: Comparison: SPD489 vs Placebo; Relationships; Test type: Superiority or Other; p = 0.1752, ANCOVA; Mean Difference (Final Values) = 7.3, 95% CI 2-sided [-3.4 to 18.0]
Statistical Analysis 5: Comparison: SPD489 vs Placebo; Total Score; Test type: Superiority or Other; p = 0.0015, ANCOVA; Mean Difference (Final Values) = 14.7, 95% CI 2-sided [5.9 to 23.6]

ADVERSE EVENTS:
Description: Safety Population defined as all subjects who took at least 1 dose of investigational product in the double-blind evaluation phase.
Arm/Group | SPD489 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/80
Other Adverse Events (participants affected / at risk) | 62/79 | 41/80
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD489 (N=79) | Placebo (N=80)
Diarrhea (Gastrointestinal disorders) | 6 | 2
Dry Mouth (Gastrointestinal disorders) | 25 | 6
Nausea (Gastrointestinal disorders) | 2 | 5
Fatigue (General disorders) | 6 | 3
Feeling Jittery (General disorders) | 10 | 0
Irritability (General disorders) | 8 | 3
Nasopharyngitis (Infections and infestations) | 4 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 1
Heart Rate Increased (Investigations) | 4 | 2
Weight Decreased (Investigations) | 8 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 0
Decreased Apetite (Metabolism and nutrition disorders) | 26 | 5
Headache (Nervous system disorders) | 20 | 2
Initial Insomnia (Psychiatric disorders) | 8 | 5
Insomnia (Psychiatric disorders) | 10 | 3
Libido Decreased (Psychiatric disorders) | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.